CLINICAL TRIAL: NCT01296646
Title: Sweet Preference and Alcohol Craving Predict Naltrexone Response in Alcoholism
Brief Title: Sweet Preference and Alcohol Craving
Acronym: SweetNal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, James Garbutt, MD, Professor of Psychiatry, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-0939; 1R21AA017503-01A2 (NIH)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Alcohol Dependence; Alcohol Abuse
Keywords: Alcohol; Alcoholics; Substance Abuse; Alcohol Abuse; Alcohol Addiction
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Naltrexone; Counseling; Practice Management, Medical; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Active Comparator): Sweet Liker, High Craver Half of this group will be on naltrexone the other half will be on placebo. All subjects will receive Brenda Therapy Sessions
  Interventions: Drug: Naltrexone; Behavioral: Brenda Therapy Sessions; Drug: Placebo
- Arm 2 (Active Comparator): Sweet Liker - Low Craver Half of this group will be on naltrexone the other half will be on placebo. All subjects will receive Brenda Therapy Sessions
  Interventions: Drug: Naltrexone; Behavioral: Brenda Therapy Sessions; Drug: Placebo
- Arm 3 (Active Comparator): Sweet Disliker - High Craver. Half of this group will be on naltrexone the other half will be on Placebo. All subjects will receive Brenda Therapy Sessions
  Interventions: Drug: Naltrexone; Behavioral: Brenda Therapy Sessions; Drug: Placebo
- Arm 4 (Active Comparator): Sweet Disliker - Low Craver; half of this group will be on naltrexone the other half on placebo. All subjects will receive Brenda Therapy Sessions
  Interventions: Drug: Naltrexone; Behavioral: Brenda Therapy Sessions; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 50 mg oral naltrexone once/day
  Other Names: Revia
Behavioral: Brenda Therapy Sessions — participants will meet with a trained therapist for nine 30-minute BRENDA therapy sessions Medical monitoring will also be conducted by study physicians and will consist of review of vital signs, concomitant medication use, and general inquiries into side effects.
  Other Names: Counselling; Therapy Sessions; Medical Management
Drug: Placebo — An inactive pill to control for non-pharmacological responses.
  Other Names: "Sugar pill"

SUMMARY:
Purpose: The proposed 2-year investigation will be the first double-blind, placebo-controlled trial examining the hedonic response to sweet taste (HRST) as a phenotypic predictor of naltrexone (NTX) response in alcohol dependence. HRST yields two primary phenotypes-Sweet Likers (SL) and Sweet Dislikers (SDL). Based on preliminary findings, HRST will be examined in conjunction with craving for alcohol to assess whether the two factors together provide a more robust predictor of NTX response. The identification of methods to predict naltrexone response in alcohol dependence is an important goal for alcohol treatment research. Currently naltrexone is not being used nearly as much as it should be, in part because clinicians do not believe it is very effective. The development of tools that would identify which patients are more likely to have a robust response to naltrexone should lead to increased use of the medication. This could help many patients who are not now having the opportunity of trying naltrexone.

There are two principal Specific Aims for the study:

Specific Aim 1. To test the hypothesis that a combination of SL/SDL status and initial alcohol craving will predict % abstinent days (%ABST) during treatment with naltrexone.

Specific Aim 2. To test whether a combination of SL/SDL status and initial alcohol craving predict % heavy drinking days (%HDD) during treatment with naltrexone.

DETAILED DESCRIPTION:
Participants: There will be 130 alcohol-dependent individuals between 18 and 65 years of age recruited to participate in this randomized placebo-controlled clinical trial. Eighty alcohol-dependent individuals will be randomized into the study and we are allowing for 50 screen failures. Participation in this study will be an alternative to standard treatment. Subjects will be blindly assessed for SL/SDL status to yield 50% representation of each trait.

Procedures (methods): Subjects who meet general inclusion/exclusion criteria based on the screening interview will complete a sweet taste assessment. Results, along with craving score, will be given to the Investigational Drug Services for randomization purposes. The study is a double-blind, randomized, placebo-controlled clinical trial in which participants will receive 50 mg oral naltrexone or matching placebo for a 12-week period. In addition participants will meet with a trained therapist for nine 30-minute BRENDA therapy sessions Medical monitoring will also be conducted by study physicians and will consist of review of vital signs, concomitant medication use, and general inquiries into side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 65 meeting DSM-IV criteria for current alcohol dependence.
2. More than 14 drinks (women) or 21 drinks (men) per week including at least 2 heavy drinking days/week on average (men > 5 drinks/day; women > 4 drinks/day) during a consecutive 30-day period within the 90 days prior to screening.
3. Ability to understand and sign written informed consent.
4. Must have a 0.0 gms/dL breathalyzer reading on the day of screening and 0.0 gms/dL on the day of randomization.
5. Must be willing to refrain from drinking for three days prior to randomization day.
6. Express a desire to achieve abstinence or to greatly reduce alcohol consumption.
7. Must have a stable residence and be able to identify an individual who could locate subject if needed.

Exclusion Criteria:

1. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., cirrhosis, unstable hypertension, seizure disorder, use of opiate medication).
2. Clinically significant psychiatric illness including: any psychotic disorder, bipolar disorder, severe depression, or suicidal ideation.
3. Other substance abuse or dependence disorder other than nicotine or alcohol.
4. Concurrent use of any psychotropic medication including antidepressants, mood stabilizers, antipsychotics, anxiolytics, stimulants, or hypnotics with the exception of stable doses of antidepressants for one month.
5. History of complicated alcohol withdrawal, i.e. withdrawal seizure or delirium tremens.
6. AST, or ALT > 3 times Upper Limit of Normal (ULN) or bilirubin > ULN.
7. Positive urine toxicology screen with the exception of cannabis. Individuals with positive cannabis screens will be excluded only if they have a history of cannabis dependence.
8. Pregnant women and women of childbearing potential who do not practice a medically acceptable form of birth control (oral or depot contraceptive, or barrier methods such as diaphragm or condom with spermicidal) and women who are breast feeding.
9. Individuals requiring inpatient treatment or more intense outpatient treatment for their alcohol dependence.
10. Participation in any clinical trial within the past 60 days.
11. Court-mandated participation in alcohol treatment or pending incarceration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Garbutt, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Garbutt JC, Kampov-Polevoy AB, Kalka-Juhl LS, Gallop RJ. Association of the Sweet-Liking Phenotype and Craving for Alcohol With the Response to Naltrexone Treatment in Alcohol Dependence: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Oct 1;73(10):1056-1063. doi: 10.1001/jamapsychiatry.2016.2157. PMID 27627782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured primarily via community advertising by radio.
Pre-assignment Details: Subjects were screened and, if met criteria, randomized to placebo or naltrexone generally within 5-10 days.
Groups:
- Placebo: Placebo taken once daily.
- Naltrexone: 50 mg of naltrexone orally daily.
Period: Overall Study
Arm/Group | Placebo | Naltrexone
Started | 40 | 40
Completed | 29 | 29
Not Completed | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naltrexone | Total
Number analyzed (Participants) | 40 | 40 | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (8.4) | 45.8 (8.6) | 47.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 28 | 29 | 57
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percent Heavy Drinking Days
Description: Percentage of heavy drinking days as derived from the Timeline Follow-back (TLFB) for the entire medication period. A heavy drinking day is defined as 5 or more standard drinks for a man and 4 or more standard drinks for a woman. A standard drink is 12-14 grams of ethanol or the amount contained in a 12 oz beer, 5 oz of wine or 1 1/2 oz of hard liquor.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 40 | 40
percentage of days
  Sweet Liker - High Craving n=9 | 0.63 (0.18) | 0.14 (0.13)
  Sweet Liker - Low Craving n=13 | 0.09 (0.12) | 0.17 (0.30)
  Sweet Disliker - High Craving n=31 | 0.19 (0.23) | 0.16 (0.20)
  Sweet Disliker - Low Craving n=27 | 0.12 (0.22) | 0.14 (0.27)

2. Secondary Outcome: Percent Days Abstinent
Description: Percentage of abstinence days as derived from the Timeline Follow-Back (TLFB) for the entire medication period.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 40 | 40
percentage of days
  Sweet Liker - High Craving n=9 | 0.27 (0.20) | 0.77 (0.29)
  Sweet Liker - Low Craving n=13 | 0.72 (0.16) | 0.67 (0.29)
  Sweet Disliker - High Craving n=31 | 0.64 (0.27) | 0.62 (0.34)
  Sweet Disliker - Low Craving n=27 | 0.61 (0.34) | 0.66 (0.27)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Subjects were asked at each visit if they had experienced any adverse events since prior visit.
Arm/Group | Placebo | Naltrexone
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/40 | 3/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Naltrexone (N=40)
Heart Attack (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Naltrexone (N=40)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No